CLINICAL TRIAL: NCT00609882
Title: Comparison of Humidified High Flow Nasal Cannula to Nasal Continuous Positive Airway Pressure for Non-Invasive Respiratory Support in Neonates
Brief Title: Comparison of Humidified High Flow Nasal Cannula to Nasal CPAP in Neonates
Acronym: HHFNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Intermountain Health Care, Inc. (Other)
Responsible Party: Bradley A. Yoder, MD, University of Utah School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24721; UofU_IRB_00024721
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Respiratory Insufficiency
Keywords: Nasal CPAP; High flow nasal cannula; Neonate
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HHFNC (Active Comparator): Infants randomized to the Humidified High Flow Nasal Cannula (HHFNC) treatment group post extubation
  Interventions: Other: Nasal CPAP; Other: Humidified High Flow Nasal Cannula (HHFNC)
- nCPAP (Active Comparator): Infants randomized to the nasal Continuous Positive Airway Pressure (nCPAP) treatment group
  Interventions: Other: Nasal CPAP; Other: Humidified High Flow Nasal Cannula (HHFNC)

INTERVENTIONS:
Other: Nasal CPAP — Infants randomized to the Standard nasal CPAP via "bubble" or ventilator support at levels of 4-8 cm H2O post extubation
Other: Humidified High Flow Nasal Cannula (HHFNC) — HHFNC

SUMMARY:
We hypothesize that the success rate for keeping babies extubated (without a breathing tube for assisted mechanical ventilation), defined as the proportion of infants remaining extubated for a minimum of 72 hours, will be equivalent among infants managed with nasal CPAP compared to humidified high flow nasal cannula (HHFNC).

DETAILED DESCRIPTION:
Respiratory failure remains a common problem in the neonatal ICU. Among premature infants with respiratory failure the use of mechanical ventilation has been associated with increased risk for secondary lung injury and subsequent development of bronchopulmonary dysplasia (BPD). As reported by Avery et al and Van Marter et al, early application of nasal continuous positive airway pressure (nCPAP) has been shown as an effective non-invasive mode of respiratory support in this population.(1, 2) Additionally, in the premature sheep and baboon models of BPD, the early use of nCPAP is accompanied by significant improvement in subsequent lung development and alveolization.(3) In light of these findings, there has been a concerted effort in most NICU's to avoid prolonged ventilator support through the early application of nCPAP.

Unfortunately, nCPAP systems are not always easily applied or tolerated in the preterm population.

Difficulties with the application of nCPAP include bulky head wraps, positional problems, compression of the nose, marked dilation and tissue breakdown of the nares, and apparent agitation, often leading to the use of potentially neurotoxic medications.(4) Previous studies have suggested that NC flows at 1-2 lpm may also generate a positive pressure in the airway of preterm infants.(5) The use of NC flow to generate positive airway pressure would minimize many of the application issues of nCPAP. However, standard NC systems used in neonates routinely employ gas that is inadequately warmed and humidified, limiting the use of such flows due to increased risk of nasal mucosa injury, and possibly increasing the risk for nosocomial infection.(4, 6) The development of humidified high flow via nasal cannulas (HHFNC) systems may obviate these problems and provide a safe, effective alternative to nCPAP in the preterm infant. Unfortunately, HHFNC does not allow the measurement of distending pressure without an invasive process such as an esophageal pressure catheter. Two recent reports have suggested that HHFNC does not provide excessive distending pressure.(7, 8) The study by Saslow and colleagues found that work of breathing and lung compliance were improved in preterm infants on HHFNC up to a maximum of 5 lpm compared to nCPAP at 6 cm H2O.(7) In comparison to nCPAP, the maximum positive distending pressure measured was 4.8 cm H2O and was not significantly increased with HHFNC flows up to 5 lpm. Kubicka and colleagues also demonstrated that the maximum distending pressure measured during support with HHFNC up to 8 lpm was < 5 cm H2O.(8)

A recent publication has suggested that HHFNC can safely and effectively be applied in the non-invasive respiratory management of premature infants with respiratory dysfunction.(9) In this retrospective analysis evaluating over 1000 infants, Shoemaker et al reported a significant decrease in ventilator days among the group of infants managed with HHFNC compared to infants previously managed with nCPAP. Additionally, they found no increased adverse effects noted such as air leak, intraventricular hemorrhage, nosocomial infection or BPD. In a smaller prospective study, Campbell et al did not find a benefit from high-flow NC among a group 40 infants < 1250 grams.(10) However, they did not use adequate humidification and the maximum "high-flow" applied was < 2 lpm. The previously noted study by Woodhead et al demonstrated that HHFNC decreased respiratory work effort and was more effective at preventing reintubation than high-flow from a standard, non-heated, non-humidified nasal cannula.(4)

Thus HHFNC, with flow rates as high as 8 lpm, is being used clinically in a large number of NICU's, including all of the units participating in this study, for management of a variety of neonatal respiratory problems. The introduction of HHFNC into clinical practice has not been accompanied by apparent changes in neonatal outcome, but this has not been systematically studied in a randomized, controlled approach.

The purpose of this randomized controlled trial is to evaluate the clinical impact of applying HHFNC to that of nCPAP among a group of infants requiring continuing non-invasive respiratory support in the NICU.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight > 1000 grams and > 27 weeks gestation
2. Candidate for non-invasive respiratory support as a result of:

   1. an intention to manage the infant with non-invasive (no endotracheal tube) respiratory support from birth initiated in the first 24 hours of life
   2. an intention to extubate an infant being managed with intubated respiratory support to non-invasive support

Exclusion Criteria:

1. Birth weight < 1000 grams
2. Estimated gestation < 29 weeks
3. Participation in a concurrent study that prohibits the use of HHFNC
4. Active air leak syndrome
5. Infants with abnormalities of the upper and lower airways; such as Pierre- Robin, Treacher-Collins, Goldenhar, choanal atresia or stenosis, cleft lip and/or palate, or
6. Infants with significant abdominal or respiratory malformations including tracheo-esophageal fistula, intestinal atresia, omphalocele, gastroschisis, and congenital diaphragmatic hernia.

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Actual)
Dates: Start 2007-12; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Compare extubation success rate, defined as % infants remaining extubated for > 72 hrs, among infants managed with HHFNC versus nCPAP | 72 hrs

SECONDARY OUTCOMES:
Compare frequency of significant apnea after extubation to HHFNC v CPAP | 7 days
Compare total duration of ventilator, positive pressure (CPAP and/or HHFNC), and oxygen use up to the time of discharge from the NICU | 3 months
Compare incidence of potential adverse effects associated with the use of nasal CPAP and HHFNC including pulmonary air leaks, nasal deformities, feeding intolerance, necrotizing enterocolitis, intestinal perforation and BPD | 3 months
Compare weight gain and the time to establish full enteral feeds (> 120 ml/kg/d) between infants on HHFNC v CPAP | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bradley A Yoder, MD, Principal Investigator — University of Utah
Locations (9):
- United States (8):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - McKay-Dee Medical Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University Hospital, Salt Lake City, Utah
  - Intermountain Medical Center, Salt Lake City, Utah
  - Dixie Medical Center, St. George, Utah
- Hebei Provincial Children's Hospital, Shijiazhuang, China

REFERENCES:
- [Background] Avery ME, Tooley WH, Keller JB, Hurd SS, Bryan MH, Cotton RB, Epstein MF, Fitzhardinge PM, Hansen CB, Hansen TN, et al. Is chronic lung disease in low birth weight infants preventable? A survey of eight centers. Pediatrics. 1987 Jan;79(1):26-30. PMID 3797169
- [Background] Van Marter LJ, Allred EN, Pagano M, Sanocka U, Parad R, Moore M, Susser M, Paneth N, Leviton A. Do clinical markers of barotrauma and oxygen toxicity explain interhospital variation in rates of chronic lung disease? The Neonatology Committee for the Developmental Network. Pediatrics. 2000 Jun;105(6):1194-201. doi: 10.1542/peds.105.6.1194. PMID 10835057
- [Background] Thomson MA, Yoder BA, Winter VT, Martin H, Catland D, Siler-Khodr TM, Coalson JJ. Treatment of immature baboons for 28 days with early nasal continuous positive airway pressure. Am J Respir Crit Care Med. 2004 May 1;169(9):1054-62. doi: 10.1164/rccm.200309-1276OC. Epub 2004 Feb 12. PMID 14962819
- [Background] Woodhead DD, Lambert DK, Clark JM, Christensen RD. Comparing two methods of delivering high-flow gas therapy by nasal cannula following endotracheal extubation: a prospective, randomized, masked, crossover trial. J Perinatol. 2006 Aug;26(8):481-5. doi: 10.1038/sj.jp.7211543. Epub 2006 May 25. PMID 16724119
- [Background] Sreenan C, Lemke RP, Hudson-Mason A, Osiovich H. High-flow nasal cannulae in the management of apnea of prematurity: a comparison with conventional nasal continuous positive airway pressure. Pediatrics. 2001 May;107(5):1081-3. doi: 10.1542/peds.107.5.1081. PMID 11331690
- [Background] Kopelman AE, Holbert D. Use of oxygen cannulas in extremely low birthweight infants is associated with mucosal trauma and bleeding, and possibly with coagulase-negative staphylococcal sepsis. J Perinatol. 2003 Mar;23(2):94-7. doi: 10.1038/sj.jp.7210865. PMID 12673256
- [Background] Saslow JG, Aghai ZH, Nakhla TA, Hart JJ, Lawrysh R, Stahl GE, Pyon KH. Work of breathing using high-flow nasal cannula in preterm infants. J Perinatol. 2006 Aug;26(8):476-80. doi: 10.1038/sj.jp.7211530. Epub 2006 May 11. PMID 16688202
- [Background] Kubicka ZJ, Limauro J, Darnall RA. Heated, humidified high-flow nasal cannula therapy: yet another way to deliver continuous positive airway pressure? Pediatrics. 2008 Jan;121(1):82-8. doi: 10.1542/peds.2007-0957. PMID 18166560
- [Background] Shoemaker MT, Pierce MR, Yoder BA, DiGeronimo RJ. High flow nasal cannula versus nasal CPAP for neonatal respiratory disease: a retrospective study. J Perinatol. 2007 Feb;27(2):85-91. doi: 10.1038/sj.jp.7211647. PMID 17262040
- [Background] Campbell DM, Shah PS, Shah V, Kelly EN. Nasal continuous positive airway pressure from high flow cannula versus Infant Flow for Preterm infants. J Perinatol. 2006 Sep;26(9):546-9. doi: 10.1038/sj.jp.7211561. Epub 2006 Jul 13. PMID 16837929
- [Derived] Yoder BA, Stoddard RA, Li M, King J, Dirnberger DR, Abbasi S. Heated, humidified high-flow nasal cannula versus nasal CPAP for respiratory support in neonates. Pediatrics. 2013 May;131(5):e1482-90. doi: 10.1542/peds.2012-2742. Epub 2013 Apr 22. PMID 23610207